CLINICAL TRIAL: NCT04034862
Title: Impact of DOlutegravir+Lamivudine Simplification on TIssue and Blood Latent Replication-competent HIV-1 Reservoirs (IDOLTIB Study)
Brief Title: Impact of DOlutegravir+Lamivudine Simplification on HIV-1 Reservoirs
Acronym: IDOLTIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gilles Darcis, Head of clinic, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13011987
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2DR (Experimental): Switch from 3 drug regimen (DTG+ABC+3TC) to 2 drug regimen (DTG+3TC)
  Interventions: Drug: Treatment simplification (dolutegravir lamivudine)
- 3DR (No Intervention): Continued 3 drug regimen treatment (DTG+ABC+3TC)

INTERVENTIONS:
Drug: Treatment simplification (dolutegravir lamivudine) — Switch from 3 drug regimen (DTG/ABC/3TC) to 2 drug regimen
  Arms: 2DR

SUMMARY:
For a few years, there has been a keen interest of clinicians and patients for "lighter" antiretroviral strategies based on two- or even single drug regimens rather than the canonical triple therapy, both as initial and maintenance therapy, despite the possibility that ongoing viral replication may occur in some patients under triple-therapy.

We will therefore propose such simplification strategy (DTG/3TC) while maintaining triple-therapy (DTG/ABC/3TC) in a control group and will perform an in depth analysis of the replication-competent reservoir in blood and in tissues as well as measurements of residual viremia and immune chronic activation/inflammation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults receiving cART for at least 2 years
* DTG/3TC/ABC as cART regimen in the previous 6 months.
* CD4 counts higher than 200 cells per μL and virological suppression for at least 2 years (plasma HIV RNA <20 copies per mL)

Exclusion Criteria:

* hepatitis C or B co-infection
* unstable liver disease
* renal impairment (estimated glomerular filtration rate <50 mL per min),
* gastrointestinal disorders that would affect the absorption of study treatment
* current use of drugs with significant interactions with dolutegravir
* current use of drugs with an impact on inflammation such as steroids.
* hospitalization for acute illness within the previous 8 weeks
* Pregnancy or breastfeeding.
* Known resistance to DTG or 3TC
* Active tuberculosis
* Anal or rectal lesions impeding rectal biopsies
* Decreased platelets count or coagulation disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The impact of dual-therapy Dolutegravir (DTG) + Lamivudine (3TC) at the level of replication-competent reservoir (RCR) in blood and in tissues. | 1 year
  Measurements of RCR in the blood and tissues (rectal biopsies)

SECONDARY OUTCOMES:
The impact of dual-therapy Dolutegravir (DTG) + Lamivudine (3TC) on residual viremia. | 1 year
The impact of dual-therapy Dolutegravir (DTG) + Lamivudine (3TC) at the level of chronic immune activation/inflammation. | 1 year
The correlation between blood and tissues RCR in a high number of patients under suppressive antiretroviral therapy. | 1 year
The level of clonal expansion in the blood and tissue RCR | 1 year
The correlation between the size of the blood/tissues RCR and the level of chronic immune activation/inflammation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Darcis, MD PhD, Principal Investigator — Liege University Hospital
Locations (1):
- Liège university hospital, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol